CLINICAL TRIAL: NCT05958199
Title: A Phase 1a/1b, Dose-Escalation/Dose-Expansion Study of NPX267 in Subjects With Solid Tumors Known to Express HHLA2/B7-H7
Brief Title: A Study of NPX267 for Subjects With Solid Tumors Known to Express HHLA2/B7-H7
Status: Suspended | Phase: Phase 1 | Type: Interventional
Why Stopped: Business decision
Sponsor: NextPoint Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NPX267-001
Record Dates: First submitted 2023-06-23; First posted 2023-07-24 (Actual); Last update posted 2025-06-27 (Actual); Status verified 2025-06

CONDITIONS: Metastatic Malignant Neoplasm
Keywords: B7-H7/HHLA2; Non-small cell lung carcinoma; renal cell carcinoma; colorectal carcinoma; cholangiocarcinoma; pancreatic cancer; urothelial carcinoma; gastric gastroesophageal carcinoma; triple negative breast carcinoma; endometrial carcinoma; cervical cancer; osteosarcoma; prostate cancer; RECIST; Dose escalation; Dose expansion
MeSH Terms: conditions — Neoplasm Metastasis; Carcinoma, Non-Small-Cell Lung; Carcinoma, Renal Cell; Colorectal Neoplasms; Cholangiocarcinoma; Pancreatic Neoplasms; Carcinoma, Transitional Cell; Triple Negative Breast Neoplasms; Endometrial Neoplasms; Uterine Cervical Neoplasms; Osteosarcoma; Prostatic Neoplasms

STUDY DESIGN:
Intervention Model Description: Dose escalation and dose expansion
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- NPX267 Treatment (Experimental)
  Interventions: Drug: NPX267

INTERVENTIONS:
Drug: NPX267 — NPX267 will be administered by intravenous infusion every three weeks until documented disease progression or participant withdrawal

SUMMARY:
NPX267 is an antibody drug targeting the inhibitory receptor for B7-H7 (HHLA2) which may control evasion of the immune response in tumors. The goal of this clinical trial is to learn whether NPX267 is safe and tolerable in patients whose cancers are known to express HHLA2 including epidermal growth factor receptor (EGFR) mutant non-small cell lung cancer. The main questions it aims to answer are:

* what is an appropriate dose to be given to patients?
* are the side effects of treatment manageable?

Participants will be evaluated for participation in the study. Patients who are treated will receive an intravenous infusion of NPX267 every three weeks if their disease has not progressed. Patients will be closely monitored by the treating physician.

DETAILED DESCRIPTION:
This trial is divided into two parts. The first part (dose escalation) will test different doses of drug to find a dose for part two. In the second part (dose expansion), more patients will be tested to see if the drug has an effect on patient's tumors.

Throughout the study, data will be collected to characterize the clinical activity of the drug. Samples of blood will be taken to help in an understanding of how the drug behaves in the body by assessing the amount of drug in the blood over time (pharmacokinetics), and changes in blood components (pharmacodynamics and safety). Tumor imaging by computed tomography (CT) or magnetic resonance imaging (MRI) will be done about every nine weeks to assess NPX267 impact on tumor growth.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed recurrent, metastatic solid tumor refractory to standard of care therapy in one of the following indications: Part 1a: non-small cell lung carcinoma (NSCLC), renal cell carcinoma (RCC), colorectal carcinoma (CRC), cholangiocarcinoma (CCA), pancreatic cancer (PDAC), urothelial carcinoma (UCC), gastric/gastroesophageal carcinoma, triple negative breast carcinoma, endometrial carcinoma, cervical cancer, osteosarcoma, and prostate cancer
* Eastern Cooperative Oncology Group (ECOG) performance status 0 or 1
* Normal bone marrow, kidney and liver function
* Willing to use highly effective contraceptive measures throughout the trial

Exclusion Criteria:

* Have any unresolved toxicity of Grade ≥ 2 from previous anti-cancer treatment, except for alopecia, chronic neuropathy > 6 months, or changes in skin pigmentation
* Have known or suspected brain metastases, unless they are clinically stable
* Known autoimmune disease requiring immunosuppressive treatment requiring the equivalent of more than 10 mg prednisone daily
* History of grade 3 immune-related pneumonitis or colitis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 131 (Estimated)
Dates: Start 2023-07-21 (Actual); Primary Completion 2025-09-20 (Estimated); Study Completion 2025-09-20 (Estimated)

PRIMARY OUTCOMES:
Incidence of dose limiting toxicity | from first dose through 21 days
  Number of subjects with dose limiting toxicity
Incidence of treatment-emergent adverse events | up to 12 weeks from first dose
  Number and type of adverse events categorized by Common Terminology Criteria for Adverse Events (CTCAE) version 5.0
Number of subjects with tumor response in tumors expressing B7-H7/HHLA2 | up to 12 weeks from first dose
  The proportion of subjects with complete or partial responses or stable disease as defined by RECIST 1.1 criteria

SECONDARY OUTCOMES:
Area under the concentration curve (AUC) of NPX267 | Following dosing on day 1, day 22, and day 43 (day 1 of 21-day treatment cycles)
  Measurement of plasma concentration over time for exposure to NPX267
Half-life in circulation (T1/2) of NPX267 | Following dosing on day 1, day 22, and day 43 (day 1 of 21-day treatment cycles)
  Measurement of the clearance of NPX267 from plasma over time
Maximum plasma concentration (Cmax) of NPX267 | Following dosing on day 1, day 22, and day 43 (day 1 of 21-day treatment cycles)
Overall survival | From first dose until death from any cause through 30 months
  Average length of survival for treated patients
Immunogenicity of NPX267 | From first dose through one year
  Number of participants with anti-drug antibodies

OTHER OUTCOMES:
Change in biomarkers of activity | From first dose through one year
  Exploratory analysis of biomarkers from collected tumor and blood samples

CONTACTS AND LOCATIONS:
Overall Officials: Leena Gandhi, MD, PhD, Study Director — NextPoint
Locations (7):
- United States (7):
  - Johns Hopkins University Sidney Kimmel Comprehensive Cancer Center, Baltimore, Maryland
  - Massachusetts General Hospital, Boston, Massachusetts
  - Albert Einstein Medical College Montefiore Medical Center, New York, New York
  - Sarah Cannon Research Institute Oncology Partners, Nashville, Tennessee
  - MD Anderson Cancer Center, Houston, Texas
  - NEXT Oncology-San Antonio, San Antonio, Texas
  - NEXT Oncology-Fairfax, Fairfax, Virginia

IPD SHARING:
Plan to Share IPD: No